CLINICAL TRIAL: NCT06313606
Title: Sparking Gut Bacteria Production of Bioactive Xenolipids in Situ
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Davis (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 2047436
Record Dates: First submitted 2023-09-23; First posted 2024-03-15 (Actual); Last update posted 2024-12-06 (Actual); Status verified 2024-12

CONDITIONS: Dietary Fat Metabolism

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dietary fat with negative control supplement (Experimental): Dietary fat-containing meal plan with a specific supplement that should not modify fat metabolism
  Interventions: Dietary Supplement: Dietary fat negative control
- Dietary fat with positive control supplement (Experimental): Dietary fat-containing meal plan with a specific supplement that may modify fat metabolism
  Interventions: Dietary Supplement: Dietary fat positive control

INTERVENTIONS:
Dietary Supplement: Dietary fat positive control — Dietary fat-containing meal plan with a specific supplement that may modify fat metabolism
  Arms: Dietary fat with positive control supplement
Dietary Supplement: Dietary fat negative control — Dietary fat-containing meal plan with a specific supplement that should not modify fat metabolism
  Arms: Dietary fat with negative control supplement

SUMMARY:
Long-chain cyclopropane fatty acids (CpFAs) are microbially-derived lipids (fats), some of which can be found in select foods and appear to be produced naturally in the gut from dietary fatty acid precursors. Some of these lipids appear to have signaling properties in the body's tissues, i.e., to help regulate cardiometabolic health. Thus, increasing the bioavailability of CpFAs in humans may have utility to improve management of blood sugar and blood lipids, or to mitigate or prevent non-alcoholic fatty liver disease (NAFLD). This study is a proof-of-principle experiment in 10 subjects, to feed dietary fats thought to enhance upper gut CpFA production. The latter will be monitored through post-meal blood and urine CpFA concentration measurements, as well as concentration in the stool.

ELIGIBILITY:
Inclusion Criteria:

* Men and women aged 18 to 50, with a Body Mass Index (BMI) categorized "normal" through "overweight" (18.5-29.9 kg/m2) and able to provide informed consent in English will be recruited to the study.

Exclusion Criteria:

* - pregnancy or lactation
* allergy or aversion to any of the foods that will be studied and/or provided
* history of gastrointestinal disorders including ulcerative colitis, Crohn's disease, celiac sprue, hereditary non-polyposis colorectal cancer (HNPCC), familial adenomatous polyposis, pancreatic disease, or liver disease
* history of any metabolic diseases (including, but not limited to: diabetes mellitus, hyperlipidemia)
* previous gastrointestinal resection or bariatric surgery
* bleeding disorders that preclude blood draws
* history of kidney disease
* recent hospital admissions (past 6 months) for heart disease (MI/CVA or CHF) or other CVD/CAD conditions under physician guided therapy
* cancer under radiation or chemotherapy treatment that is active or within 6 months of treatment
* regular alcohol intake of > 2 drinks/day (equivalent to 720 mL of beer, 240 mL of wine, or 90 mL of spirits) and unwilling to abstain during the run-in week and test day
* use of tobacco and/or marijuana, hookahs, e-cigarettes (e-cigs, vapes, etc.) and not willing to abstain during the run-in week and test day
* use of illicit drugs and not willing to abstain during the run-in week and test day
* BMI greater than 30 kg/m2 or below 18.5 kg/m2
* regular (daily to weekly) use of over the counter (OTC) weight-loss aids, anti-acids or anti-inflammatories, and unwilling or unable to stop taking during the run-in week and test day
* regular OTC dietary supplements that interfere with the test foods being studied including pills, chewables, liquids or powders for the following: fiber, fish oil (including cod liver oil), probiotics, and unwilling or unable to stop taking during the run-in week and test day
* oral or IV antibiotic use in the past 6 months (could defer participation until 6 months post-completion of course of antibiotics)
* seated blood pressure >140/90 mmHg
* fasting clinical lab tests outside acceptable values as ascertained at the screening blood draw
* current use of specific prescription medication(s) that could impact gut physiology, gut microbiota, or other systems relevant to metabolism and fat PK
* inability to freely give informed consent in English

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Estimated)
Dates: Start 2024-04-01 (Actual); Primary Completion 2025-05-31 (Estimated); Study Completion 2025-05-31 (Estimated)

PRIMARY OUTCOMES:
Cyclopropane fatty acid metabolite concentrations in blood, urine, and stool | 24-48 hours following test meal intake
  Change in blood, urine, or gastrointestinal (stool) CpFA fatty acids following dietary fat intake

CONTACTS AND LOCATIONS:
Overall Officials: Sean H. Adams, PhD, Principal Investigator — University of California, Davis
Locations (1):
- University of California, Davis School of Medicine, Sacramento, California, United States

IPD SHARING:
Plan to Share IPD: No